CLINICAL TRIAL: NCT06277258
Title: Outcome of "Patient Empowerment" in the Management of Gestational Diabetes Mellitus: A Clustered Randomized Controlled Trial
Brief Title: Patient Empowerment in the Management of Gestational Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Public Health Foundation of Bangladesh (Other)
Responsible Party: Principal Investigator, Tabassum Parveen, Member, Public Health Foundation of Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BSMMU/2022/9656
Record Dates: First submitted 2022-12-15; First posted 2024-02-26 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus in Pregnancy
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: At the end of the study, the outcome will be assessed by blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Empowerment Model (Experimental): Patients will be empowered to manage gestational diabetes mellitus themselves by acquiring knowledge and skill to monitor blood sugar levels, adjusting meals and daily activities.
  Interventions: Other: Patient Empowerment model
- Standard of care (No Intervention): Patients will get the conventional way of management where patients get advice about a diet chart with a fixed menu and injection of insulin to control blood sugar levels.

INTERVENTIONS:
Other: Patient Empowerment model — Session I
  * Knowledge about the disease, calories & diet distribution, physical activities, symptoms of hypoglycemia, Blood Glucose target etc.
  * Training on use of glucometer and record keeping Session II
  * Evaluation and interpretation of sugar level based on the sugar chart.
  * Tuning of diet and exercise if needed.
  * Discussion about the challenges faced by the patient during maintenance of sugar level.
  Session III & ongoing
  * Tuning of the diet based on calories, evaluation of the understanding
  * Assessment of patient satisfaction
  * Assessment of patients' knowledge and skill to designate her as "Empowered"
  Assurance and counseling of patient and family will be rendered in each session.
  Arms: Patient Empowerment Model

SUMMARY:
This study is a clustered randomized controlled trial assessing the outcome of "Patient Empowerment" in the management of Gestational Diabetes Mellitus by applying the patient empowering model in the intervention group and the conventional method of treatment in the control group. It will be conducted in four centres in Dhaka city of Bangladesh. The primary outcome measures will be determining the frequency of good fetomaternal and neonatal outcome through glycemic control. Target of Glycemic Status: For Pregnant Mother, Fasting, 95 mg/dL (5.3 mmol/L), Two-hour postprandial,120 mg/dL (6.7 mmol/L), For Neonate glycemic status at or above 2.5 mmol/l. Maternal outcome during pregnancy - Decrease chance of antenatal infections that is Vulvovaginitis and recurrent UTI, Decrease pre-eclampsia, Decrease Antepartum Hemorrhage and Polyhydramnios. Maternal outcome in the form of mode of safe delivery- Increase frequency of vaginal delivery, Decrease chance of obstructed labour. Maternal outcome after delivery- Decrease chance of Postpartum Hemorrhage, Decrease chance of puerperal sepsis. Fetal Outcome- Less chance of Intra uterine death and prematurity. Neonatal Outcome- Less chance of Birth injury, Birth asphyxia, Perinatal death, Good Apgar score (≥ 7) in 1st and 5th minute, Less need for NICU care and Less chance of macrosomia (≥ 4 kg) at term. Fewer proportion of patients will require insulin to manage GDM. The secondary outcomes will be patient satisfaction and the patient will be a future resource person.

DETAILED DESCRIPTION:
Procedure of Study (Including methods of intervention, measurement, estimation etc.):

Screen positive GDM patients will be recruited according to inclusion and exclusion criteria. After taking consent they will be registered for study purpose. According to computer generated randomization the health centres will be allocated and single method of management either patient empowerment or conventional method will be adopted for the whole cluster of the respective health centre. The intervention group will only receive the "Patient Empowerment' package.

The patients of intervention group, along with antenatal check-up, will go through the first session of the empowerment package on the first day of recruitment. Then they will be evaluated through structured questions to know their level of perception/ understanding and retention about the diabetes and its management. Those who will perform to get at least 80% out of 100 will be recognized as empowered. Who fail to achieve that they will be called for next seating. Patients unwilling to go through the process or failed to achieve the targeted score within three seating will be excluded. Those who fulfilled the target, they will be advised to follow the calorie and diet distribution schedule. They will be advised to return back 2 days later, with the blood sugar chart (6 times per day) by SMBG (Self-monitoring of blood glucose). The respondents will get the materials like measuring cup, hand manuals on diabetes, glucometer and chart for record keeping.

After evaluating the sugar chart, if they are found poor performer they will be counselled and trained further and will have to come back again after two days. At the same time patient's satisfaction will be assessed with LIKERT scale. Frequency of further visit will depend on patient's performance.

All the respondents from both groups are supposed to come for ANC at least at monthly interval initially up to 28 weeks and then fortnightly up to 36 weeks and then weekly up to delivery; frequency of the visit may be more if necessary. For Conventional (non- intervention) group at least 2 to 3 times blood sugar level should be checked within the follow up period. Then all the pertinent variables will be recorded, analyzed as per study objective and outcome, to evaluate the effectiveness of patient empowerment in the management of GDM.

Blood sample collection:

Patients of GDM will be trained to measure their own blood sugar level (both fasting and 2 hours' postprandial) by Glucometer at home and to maintain a blood sugar chart.

Laboratory methods:

In this study design apart from routine antenatal screening tests no other additional laboratory investigation will be done unless be otherwise needed on medical ground.

Follow up of the patients:

Both the study group and comparison group will be followed up as per study protocol at monthly interval initially up to 28 weeks and then fortnightly up to 36 weeks and then weekly up to delivery; frequency of the visit may be more if necessary.

Data Collection Tools:

Pre-tested semi structured questionnaire/interview schedule and checklist.

Data Collection Procedure:

GDM cases will be enrolled in this study with taking written consent on the consent form. Data will be collected by multiple techniques like face to face interview, records, findings of physical examination and observation, information on concerned variables and will be documented. Among the variables the fasting blood sugar and 2 hours after ingestion of 75-gram glucose will be considered as baseline for detection of GDM as screening test between 14 to 34 weeks of gestation. Patient empowerment

All the clinical and investigative findings and therapeutic variables will be documented during each antenatal visit. The ANC and its frequency should be according to conventional schedule (Monthly up to 28 weeks, fortnightly up to 36 weeks and then weekly up to delivery in low risk cases and for high risk the frequency of visit will be more). In both the groups from patient's blood sugar chart, average blood sugar value will be documented monthly. Each patient will be followed up to the end of puerperium that is 6 weeks after delivery.

From each institute, data will be collected with separate registration name and number and will be stored separately.

Statistical analysis:

The data will be analyzed according to cluster randomized trial protocol; and all statistical analysis will be based on Intention to Treat (ITT) approach. Descriptive statistics will be generated for all base line and follow-up data (frequency and relative frequency for categorical data, means with standard deviations (SDs) or 95% confidence intervals (CIs) for normally distributed continuous data and for non-normal data median and interquartile ranges.

Univariable associations between baseline patient characteristics and outcome will be assessed using univariable Cox regression. All statistically significant predictors will be assessed for possible confounding. Potential confounders measured at baseline will be selected based on a directed acyclic graph (DAG) and univariate association finding. Tests based on Schoenfeld residuals will be used to identify violations of the proportional hazards assumption. Impact of intervention on for primary outcome (adverse pregnancy outcome) will be assessed using multilevel cox proportional hazard regression adjusting for plausible confounders. Multilevel modelling will include a shared frailty term in the model to account for hospital-level clustering. The between-group differences will be assessed enabling simultaneous examination of cluster and individual-level influences on outcomes. Adjustment of the result for between-cluster variation will thus be achieved. The effects of the intervention on maternal and neonatal outcomes and changes in physical activity and diet will be analysed by using generalized linear latent and mixed models and multilevel mixed-effects linear regression by fitting random effects models. All analysis will be performed in Stata S/E version 17.

Quality assurance strategy:

From research team, PI, Co-PI and other investigators and local GOB health managers will work together for effective implementation, monitoring and evaluation of interventions. They will jointly monitor the progress and oversee any deviation from the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Screen positive GDM cases, who have not been managed for diabetes by any means
2. Gestational age from18 weeks to 36 weeks

Exclusion Criteria:

1. Known history of diabetes before pregnancy
2. Women with twin or multiple pregnancies

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 459 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-11-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants with adverse maternal pregnancy outcome | Monthly from enrolment day up to 28 weeks of gestation, fortnightly from 28 weeks to 36 weeks of gestation, weekly from 36 weeks of gestation up to delivery, during delivery, Within 24 hours of delivery, 1 week, 2 weeks & 6 weeks of delivery
  Maternal pregnancy outcome are antenatal infection, Preeclampsia, polyhydramnios, Ante and post partum Haemorrhage, Puerperal sepsis. Maternal death.
Number of Participants with adverse foetal outcome | During delivery, After delivery- within 24 hours
  Adverse foetal outcome include prematurity, Birth injury, Birth asphyxia, Perinatal death, NICU admission macrosomia (≥ 4 kg) at term, hypoglycaemia (≤ 2.5 mmol/l)
Number of Participants with adequate glycaemic control | Monthly from enrollment day upto 28 weeks of gestation, fortnightly from 28 weeks to 36 weeks of gestation, weekly from 36 weeks of gestation upto delivery
  Adequate glycaemic control include (a) 80% of blood glucose reading of the month with in normal range. (b) No requirement of insulin or pharmacological agents to manage GDM,

SECONDARY OUTCOMES:
Maternal satisfaction | Monthly from enrollment day upto 28 weeks of gestation, fortnightly from 28 weeks to 36 weeks of gestation, weekly from 36 weeks of gestation upto delivery, during delivery, Within 24 hours of delivery, 1 week, 2 weeks & 6 weeks of delivery
  Patient satisfaction will be assessed through the LIKERT rating scale ranging from strongly satisfied to strongly dissatisfied. The maximum value is 5 which means the patient is strongly satisfied with the service and the minimum value is 1 wchich means the patient is strongly dissatisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Tabassum Parveen, FCPS, Principal Investigator — Professor, Department of Fetomaternal Medicine, BSMMU
Locations (3):
- Bangladesh (3):
  - Azimpur Maternity hospital ( MCHTI), Dhaka
  - Shaheed Suhrawardy Medical College (ShSMC), Dhaka
  - Bangabandhu Sheikh Mujib Medical University (BSMMU), Dhaka

IPD SHARING:
Plan to Share IPD: No
No plan of data sharing before completion of study, if required then will be done with the prior permission of the funding agency

REFERENCES:
- [Background] Diagnostic Criteria and Classification of Hyperglycaemia First Detected in Pregnancy. Geneva: World Health Organization; 2013. Available from http://www.ncbi.nlm.nih.gov/books/NBK169024/ PMID 24199271
- [Background] Biswas A, Dalal K, Abdullah ASM, Rahman AKMF, Halim A. Gestational Diabetes: Exploring the Perceptions, Practices and Barriers of the Community and Healthcare Providers in Rural Bangladesh: A Qualitative Study. Diabetes Metab Syndr Obes. 2020 Apr 23;13:1339-1348. doi: 10.2147/DMSO.S238523. eCollection 2020. PMID 32425566
- [Background] Rieck S, Kaestner KH. Expansion of beta-cell mass in response to pregnancy. Trends Endocrinol Metab. 2010 Mar;21(3):151-8. doi: 10.1016/j.tem.2009.11.001. Epub 2009 Dec 16. PMID 20015659
- [Background] Muche AA, Olayemi OO, Gete YK. Effects of gestational diabetes mellitus on risk of adverse maternal outcomes: a prospective cohort study in Northwest Ethiopia. BMC Pregnancy Childbirth. 2020 Feb 3;20(1):73. doi: 10.1186/s12884-020-2759-8. PMID 32013909
- [Background] Zhuang W, Lv J, Liang Q, Chen W, Zhang S, Sun X. Adverse effects of gestational diabetes-related risk factors on pregnancy outcomes and intervention measures. Exp Ther Med. 2020 Oct;20(4):3361-3367. doi: 10.3892/etm.2020.9050. Epub 2020 Jul 27. PMID 32855709
- [Background] Martis R, Crowther CA, Shepherd E, Alsweiler J, Downie MR, Brown J. Treatments for women with gestational diabetes mellitus: an overview of Cochrane systematic reviews. Cochrane Database Syst Rev. 2018 Aug 14;8(8):CD012327. doi: 10.1002/14651858.CD012327.pub2. PMID 30103263
- [Background] Crowther CA, Hiller JE, Moss JR, McPhee AJ, Jeffries WS, Robinson JS; Australian Carbohydrate Intolerance Study in Pregnant Women (ACHOIS) Trial Group. Effect of treatment of gestational diabetes mellitus on pregnancy outcomes. N Engl J Med. 2005 Jun 16;352(24):2477-86. doi: 10.1056/NEJMoa042973. Epub 2005 Jun 12. PMID 15951574
- [Background] Moreno-Castilla C, Mauricio D, Hernandez M. Role of Medical Nutrition Therapy in the Management of Gestational Diabetes Mellitus. Curr Diab Rep. 2016 Apr;16(4):22. doi: 10.1007/s11892-016-0717-7. PMID 26879305
- [Background] Luczynski W, Glowinska-Olszewska B, Bossowski A. Empowerment in the Treatment of Diabetes and Obesity. J Diabetes Res. 2016;2016:5671492. doi: 10.1155/2016/5671492. Epub 2016 Dec 20. PMID 28090541
- [Background] American Diabetes Association. 2. Classification and Diagnosis of Diabetes: Standards of Medical Care in Diabetes-2021. Diabetes Care. 2021 Jan;44(Suppl 1):S15-S33. doi: 10.2337/dc21-S002. PMID 33298413
- [Background] International Association of Diabetes and Pregnancy Study Groups Consensus Panel; Metzger BE, Gabbe SG, Persson B, Buchanan TA, Catalano PA, Damm P, Dyer AR, Leiva Ad, Hod M, Kitzmiler JL, Lowe LP, McIntyre HD, Oats JJ, Omori Y, Schmidt MI. International association of diabetes and pregnancy study groups recommendations on the diagnosis and classification of hyperglycemia in pregnancy. Diabetes Care. 2010 Mar;33(3):676-82. doi: 10.2337/dc09-1848. No abstract available. PMID 20190296
- [Background] Bener A, Saleh NM, Al-Hamaq A. Prevalence of gestational diabetes and associated maternal and neonatal complications in a fast-developing community: global comparisons. Int J Womens Health. 2011;3:367-73. doi: 10.2147/IJWH.S26094. Epub 2011 Nov 7. PMID 22140323
- [Background] Kim SY, Saraiva C, Curtis M, Wilson HG, Troyan J, Sharma AJ. Fraction of gestational diabetes mellitus attributable to overweight and obesity by race/ethnicity, California, 2007-2009. Am J Public Health. 2013 Oct;103(10):e65-72. doi: 10.2105/AJPH.2013.301469. Epub 2013 Aug 15. PMID 23947320
- [Background] Gupta Y, Kalra B, Baruah MP, Singla R, Kalra S. Updated guidelines on screening for gestational diabetes. Int J Womens Health. 2015 May 19;7:539-50. doi: 10.2147/IJWH.S82046. eCollection 2015. PMID 26056493
- [Background] Agarwal MM. Gestational diabetes mellitus: An update on the current international diagnostic criteria. World J Diabetes. 2015 Jun 25;6(6):782-91. doi: 10.4239/wjd.v6.i6.782. PMID 26131321
- [Background] HAPO Study Cooperative Research Group. Hyperglycemia and Adverse Pregnancy Outcome (HAPO) Study: associations with neonatal anthropometrics. Diabetes. 2009 Feb;58(2):453-9. doi: 10.2337/db08-1112. Epub 2008 Nov 14. PMID 19011170
- [Background] Herath H, Herath R, Wickremasinghe R. Gestational diabetes mellitus and risk of type 2 diabetes 10 years after the index pregnancy in Sri Lankan women-A community based retrospective cohort study. PLoS One. 2017 Jun 23;12(6):e0179647. doi: 10.1371/journal.pone.0179647. eCollection 2017. PMID 28644881
- [Background] O'Kane MJ, Pickup J. Self-monitoring of blood glucose in diabetes: is it worth it? Ann Clin Biochem. 2009 Jul;46(Pt 4):273-82. doi: 10.1258/acb.2009.009011. Epub 2009 May 19. PMID 19454538
- [Background] Reader DM. Medical nutrition therapy and lifestyle interventions. Diabetes Care. 2007 Jul;30 Suppl 2:S188-93. doi: 10.2337/dc07-s214. PMID 17596470
- [Background] Carolan-OIah MC. Educational and intervention programmes for gestational diabetes mellitus (GDM) management: An integrative review. Collegian. 2016;23(1):103-14. doi: 10.1016/j.colegn.2015.01.001. PMID 27188046
- [Background] Mohebbi B, Tol A, Sadeghi R, Mohtarami SF, Shamshiri A. Self-management Intervention Program Based on the Health Belief Model (HBM) among Women with Gestational Diabetes Mellitus: A Quazi-Experimental Study. Arch Iran Med. 2019 Apr 1;22(4):168-173. PMID 31126174
- [Background] Boutati EI, Raptis SA. Self-monitoring of blood glucose as part of the integral care of type 2 diabetes. Diabetes Care. 2009 Nov;32 Suppl 2(Suppl 2):S205-10. doi: 10.2337/dc09-S312. PMID 19875553
- [Background] Jovanovic L, Pettitt DJ. Treatment with insulin and its analogs in pregnancies complicated by diabetes. Diabetes Care. 2007 Jul;30 Suppl 2:S220-4. doi: 10.2337/dc07-s220. No abstract available. PMID 17596476
- [Background] Lapolla A, Dalfra MG, Fedele D. Insulin therapy in pregnancy complicated by diabetes: are insulin analogs a new tool? Diabetes Metab Res Rev. 2005 May-Jun;21(3):241-52. doi: 10.1002/dmrr.551. PMID 15818714
- [Background] Wei Y, Yang H, Zhu W, Hod M, Hadar E. Adverse pregnancy outcome among women with pre-gestational diabetes mellitus: a population-based multi-centric study in Beijing. J Matern Fetal Neonatal Med. 2017 Oct;30(20):2395-2397. doi: 10.1080/14767058.2016.1250257. Epub 2016 Nov 8. PMID 27822972
- [Background] Zheng Y, Shen Y, Jiang S, Ma X, Hu J, Li C, Huang Y, Teng Y, Bao Y, Zhou J, Hu G, Tao M. Maternal glycemic parameters and adverse pregnancy outcomes among high-risk pregnant women. BMJ Open Diabetes Res Care. 2019 Nov 13;7(1):e000774. doi: 10.1136/bmjdrc-2019-000774. eCollection 2019. PMID 31798901
- [Background] Bashir M, Baagar K, Naem E, Elkhatib F, Alshaybani N, Konje JC, Abou-Samra AB. Pregnancy outcomes of early detected gestational diabetes: a retrospective comparison cohort study, Qatar. BMJ Open. 2019 Feb 19;9(2):e023612. doi: 10.1136/bmjopen-2018-023612. PMID 30782883